CLINICAL TRIAL: NCT00585494
Title: Prevalence of Inpatient Hyperglycemia: Risks, Complications and Outcomes
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2007-0199
Record Dates: First submitted 2007-12-27; First posted 2008-01-03 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preoperative orthopedic: Patients undergoing elective total hip, knee and spinal surgery at University of Wisconsin hospital, having their preoperative visit between December 1, 2007 and November 30, 2008.

SUMMARY:
This protocol will determine the prevalence of hyperglycemia and diabetes in the elective orthopedic population at the University of Wisconsin. It will also determine if there is a difference in outcomes. The study hypothesizes that at least 10% of patients will have some degree of impaired glucose regulation that has previously been undiagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Undergoing elective total knee, hip or lumbar spinal surgery

Exclusion Criteria:

* Pregnancy
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University of Wisconsin orthopedic clinic patients ages 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Sheehy, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Sheehy AM, Benca J, Glinberg SL, Li Z, Nautiyal A, Anderson PA, Squire MW, Coursin DB. Preoperative "NPO" as an opportunity for diabetes screening. J Hosp Med. 2012 Oct;7(8):611-6. doi: 10.1002/jhm.1958. Epub 2012 Aug 7. PMID 22887757

RESULTS

PARTICIPANT FLOW:
Groups:
- Preoperative Orthopedic: Patients undergoing elective total hip, knee and spinal surgery at UW hospital, having their preoperative visit between December 1, 2007 and November 30, 2008.
Period: Overall Study
Arm/Group | Preoperative Orthopedic
Started | 300
Completed | 244
Not Completed | 56

BASELINE CHARACTERISTICS:
Arm/Group | Preoperative Orthopedic
Number analyzed (Participants) | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 197
  >=65 years | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 134
Region of Enrollment [Number; unit: participants]
  United States | 302

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Hyperglycemia in the Elective Orthopedic Population
Description: Number of orthopedic patients that have elevated fasting blood glucose levels preoperatively
Time Frame: 1 year
Measure: Number; unit: patients
Arm/Group | Preoperative Orthopedic
Number analyzed (Participants) | 244
patients | 140

2. Secondary Outcome: Prevalence of Undiagnosed Diabetes in the Elective Orthopedic Population.
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Prevalence of Adverse Outcomes in the Hyperglycemic Elective Orthopedic Population.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Preoperative Orthopedic
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes